CLINICAL TRIAL: NCT05872724
Title: Clinical Study on Optimization of Postoperative Adjuvant Therapy for Cervical Cancer Based on MRD
Brief Title: Optimization of Postoperative Adjuvant Therapy for Cervical Cancer Based on MRD(Minimal Residual Disease)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, jing xue, Associate chief physician, Suzhou Municipal Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Optimize
Record Dates: First submitted 2023-04-12; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Chemoradiotherapy; Chemotherapy, Adjuvant; zimberelimab

STUDY DESIGN:
Intervention Model Description: cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Eligible subjects were assigned to high-risk or medium-risk groups based on Peter's criteria and Sedlis criteria. Patients with a high-risk classification or MRDc0 (+) status received a treatment consisting of conventional pelvic concurrent chemoradiotherapy, adjuvant chemotherapy, four courses of immunotherapy, continued immunotherapy with MRDIn(+), and follow-up monitoring with MRDIn(-)
  Interventions: Drug: Chemoradiotherapy + Adjuvant chemotherapy and Zimberelimab
- Arm B (Experimental): Patients deemed intermediate risk and with MRDc0 (-) status received concurrent chemoradiotherapy in the small pelvic target volume, four courses of immunotherapy, continued immunotherapy with MRDIn(+), and follow-up monitoring with MRDIn(-)
  Interventions: Drug: Chemoradiotherapy (small pelvic) + Zimberelimab

INTERVENTIONS:
Drug: Chemoradiotherapy + Adjuvant chemotherapy and Zimberelimab — * Radiation therapy:
    1. Irradiation mode and dose: 6MV-X-ray (6Megavoltage-X-ray), IMRT or RapidArc-IMRT were used for external radiotherapy. External radiotherapy dose: PTV (Planning Target Volume) 45-50Gy/25 times.
  * Chemotherapy:
    1. Concurrent chemotherapy: Cisplatin monotherapy: DDP 75 mg/m2 for 3 days, q3w. Carboplatin or nedaplatin may be used in patients that cannot tolerate cisplatin.
    2. Adjuvant chemotherapy: After the concurrent chemoradiotherapy, 4 cycles of consolidation chemotherapy plus immunotherapy are recommended for patients with high risk or MRDc0 (+). Recommended chemotherapy regimen: liposome paclitaxel 135mg/m2 d1 +DDP 25 mg/m2 D1-3, Q21.
  * Zimberelimab injection:
    240 mg, IV, q3w. Start the drug one day before the start of postoperative radiotherapy.
  Arms: Arm A
Drug: Chemoradiotherapy (small pelvic) + Zimberelimab — Radiation therapy:
  1. Target volume of radiotherapy for small pelvis: CTVp includes tumor bed area, paracentral area and part of vagina; CTVn includes bilateral internal iliac, external iliac and obturator lymphatic drainage areas. Upper boundary to sacroiliac joint level, lower boundary to 2cm below vaginal stump.
  Chemotherapy:
  Concurrent chemotherapy: Cisplatin monotherapy: DDP 75 mg/m2 for 3 days, q3w. Carboplatin or nedaplatin may be used in patients that cannot tolerate cisplatin.
  Adjuvant chemotherapy: After the concurrent chemoradiotherapy, 4 cycles of adjuvant immunotherapy are recommended for patients in good general condition (ECOG: 0-1) with medium risk and MRDc0 (-).
  Zimberelimab injection: 240 mg, IV, q3w. Start the drug one day before the start of posterior radiotherapy.
  Arms: Arm B

SUMMARY:
This study is a prospective cohort clinical trial that aims to investigate the safety and efficacy of a combined chemoradiotherapy and immunotherapy treatment for early postoperative cervical cancer. Specifically, this study seeks to evaluate the ability of MRD-based screening to detect and monitor changes in MRD status at different stages of treatment, its potential for use in monitoring patient recurrence rates and in prognosis evaluation. In addition, this study will investigate the safety and effectiveness of chemoradiotherapy combined with immunotherapy as a postoperative adjuvant therapy for patients identified to be at risk of early cervical cancer based on MRD screening.

DETAILED DESCRIPTION:
The study comprised of three periods; a screening period (within 28 days prior to informed consent), a treatment period (defined as the time from the initiation of treatment to its termination for any reason), and a follow-up period (consisting of end-of-treatment visits, safety visits, and survival follow-up). During the screening period, participants underwent eligibility evaluations, including tissue and blood sample collection for biomarker detection. Eligible subjects were divided into high-risk and intermediate-risk groups based on Peter's criteria and Sedlis criteria, with patients in the high-risk group or those identified as MRDc0 (+) (3 days after surgery to 10 days before adjuvant therapy) receiving conventional pelvic concurrent chemoradiotherapy, adjuvant chemotherapy, and four courses of immunotherapy. Patients in the intermediate-risk group and those identified as MRDc0 (-) received simultaneous chemoradiotherapy in the target volume of the small pelvis, four courses of immunotherapy, continued immunotherapy with MRDIn(+)(2 months after initiation of immunotherapy), and follow-up monitoring with MRDIn(-). Subjects returned to the hospital for a safety follow-up 28 days (±7d) after the last dose to track the outcome of adverse events. Safety visits consisted of vital sign measurements, laboratory tests, and other protocol-required assessments to evaluate adverse events, concomitant medications, and concomitant therapy. At the end of treatment, subjects began survival follow-up every 3 months (±7d). Radiographic assessments were conducted at this frequency until disease progression, death, loss of follow-up, withdrawal of informed consent, initiation of follow-up antitumor therapy, or investigator-initiated termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathological and clinical (FIGO 2018) stage ⅠB2 ~II A2 cervical cancer.
2. Above the age of 18.
3. General status: ECOG score 0-2.
4. Be able to understand the research scheme, voluntarily participate in the study, and sign the informed consent.
5. Good compliance, able to cooperate with the collection of specimens at each node and provide corresponding clinical information.

Exclusion Criteria:

1. Suffering from other malignant tumors.
2. Do not receive the specified treatment or change the treatment regimen before the disease progresses.
3. The study cannot be followed up according to the defined clinical follow-up period.
4. Unable to accept or provide CT or other designated therapeutic evaluation means.
5. Have an autoimmune disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2028-01-16 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
3-year DFS in ITT population (intent-to-treat population) | 3-year
  DFS (disease-free survival) is the time between the start of enrollment and the recurrence of disease, or death from any cause.

SECONDARY OUTCOMES:
3-year DFS with different MRD status and changes | 3-year
  DFS (disease-free survival) is the time between the start of enrollment and the recurrence of disease, or death from any cause
2-year DFS with different MRD status and changes | 2-year
  DFS (disease-free survival) is the time between the start of enrollment and the recurrence of disease, or death from any cause
1-year DFS with different MRD status and changes | 1-year
  DFS (disease-free survival) is the time between the start of enrollment and the recurrence of disease, or death from any cause
3-year OS rates in patients with different MRD status and changes | 3-year
  OS (overall survival) is the overall time from enrollment to death from any cause
AE | Up to 28 days after the end of treatment
  Adverse events (AE) were determined and graded according to NCI CTC AE 5.0, Collect the incidence of adverse events (AEs), the incidence of serious adverse events (SAEs), the incidence of CTCAE grade 3 or above (rated based on CTCAE 5.0), the correlation of adverse events, actions taken and outcomes, etc.

OTHER OUTCOMES:
Disease recurrence based on MRD monitoring methods | through study completion, an average of 3-6 months
  The time from MRD(-) to MRD(+)
Negative conversion rate of MRD (+) patients after intensive adjuvant therapy | through study completion, an average of 3-6 months
  Incidence of conversion from MRD(+) to MRD(-) after adjuvant therapy
To explore the correlations of genes detected by next-generation sequencing, MRI-based response patterns and biomarkers of peripheral blood with the efficacy of treatment. | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: jing xue, Principal Investigator — The Affiliated Suzhou Hospital of Nanjing Medical University
Locations (1):
- The Affiliated Suzhou Hospital of Nanjing Medical University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
CRF (Case Report Form) and ICF (Informed Consent Form) will be shared in the future